CLINICAL TRIAL: NCT06299761
Title: An Open-Label, Multicenter, First-in-Human, Dose-Escalation and Dose-Expansion, Phase 1/2 Study of BBI-825 and BBI-825 in Combination With Select Targeted Therapies in Subjects With Locally Advanced or Metastatic Solid Tumors With Resistance Gene Amplifications
Brief Title: Study of the RNR Inhibitor BBI-825 in Subjects With Tumors With Resistance Gene Amplifications
Acronym: STARMAP
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Strategic decision made following an assessment of preliminary PK data from the Part 1 portion of the trial showing a lack of dose proportional exposure and the increasing complexity and associated development costs in this landscape.
Sponsor: Boundless Bio (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BBI-825-101
Record Dates: First submitted 2024-02-26; First posted 2024-03-08 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Solid Tumor
Keywords: Amplification; Oncogene Amplification; ribonucleotide reductase inhibitor; RNR inhibitor

STUDY DESIGN:
Intervention Model Description: BBI-825 single agent dose escalation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single Agent Dose Escalation (Experimental): Single agent BBI-825, administered orally, twice daily, in 28-day cycles
  Interventions: Drug: BBI-825

INTERVENTIONS:
Drug: BBI-825 — Oral RNR inhibitor
  Other Names: ribonucleotide reductase inhibitor

SUMMARY:
BBI-825 is a potent, selective, oral, small molecule inhibitor of ribonucleotide reductase (RNR). This is a first-in-human, open-label, non-randomized, 3-part, Phase 1/2 study to determine the safety profile and identify the maximum tolerated dose and recommended Phase 2 dose of BBI-825 administered as a single agent and in combination with select targeted therapies.

DETAILED DESCRIPTION:
BBI-825 will be administered orally (PO) twice daily (BID) to subjects with locally advanced or metastatic non-resectable solid tumors, whose disease has progressed despite all standard therapies or for whom no further standard or clinically acceptable therapy exists.

ELIGIBILITY:
Inclusion Criteria:

* Locally advanced or metastatic non-resectable solid tumors, whose disease has progressed despite all standard therapies or for whom no further standard or clinically acceptable therapy exists,
* Availability of FFPE tumor tissue, archival or newly obtained,
* Measurable disease as defined by RECIST Version 1.1,
* Adequate hematologic function,
* Adequate hepatic and renal function,
* Eastern Cooperative Oncology Group performance status (ECOG PS) 0 or 1,
* Other inclusion criteria per study protocol.

Exclusion Criteria:

* Prior exposure to a selective RNR inhibitor (Note: Prior exposure to chemotherapies with nonselective RNR inhibitory activity e.g., gemcitabine is permitted),
* Receipt of any approved or considered standard of care anticancer drug(s) or biological product(s) within 4 weeks or 5 half-lives,
* Hematologic malignancies,
* Primary CNS malignancy, leptomeningeal disease, or symptomatic active CNS metastases, with exceptions per study protocol,
* Prior or concurrent malignancies, with exceptions per study protocol,
* History of HBV, HCV, or HIV infection,
* Clinically significant cardiac condition,
* Active or history of interstitial lung disease (ILD) or pneumonitis, or history of ILD or pneumonitis requiring steroids or other immunosuppressive medications,
* QTcF > 470 msec,
* Concurrent use of strong inhibitors or inducers of CYP3A, CYP2C8, CYP2C9, or CYP2C19,
* Other exclusion criteria per study protocol.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2024-03-28 (Actual); Primary Completion 2025-06-25 (Actual); Study Completion 2025-06-25 (Actual)

PRIMARY OUTCOMES:
Frequency and severity of treatment emergent adverse events (TEAEs) of BBI-825 | Start of Cycle 1 until 30 days following last dose (each cycle is 28 days)
  TEAEs will be assessed and severity assigned by using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), version 5.0.
Maximum Tolerated Dose (MTD) and/or Recommended Phase 2 Dose (RP2D) of BBI-825 | Start of Cycle 1 until 30 days following last dose (each cycle is 28 days)
  The MTD and/or RP2D of BBI-825 will be determined.

SECONDARY OUTCOMES:
Maximum observed plasma concentration (Cmax) of BBI-825 | Start of Cycle 1 until Day 1 of last treatment cycle (each cycle is 28 days)
  Maximum observed plasma concentration (Cmax) of BBI-825 will be determined.
Trough observed plasma concentration (Ctrough) of BBI-825 | Start of Cycle 1 until Day 1 of last treatment cycle (each cycle is 28 days)
  Trough observed plasma concentration (Ctrough) of BBI-825 will be determined.
Time to Cmax (Tmax) of BBI-825 | Start of Cycle 1 until Day 1 of last treatment cycle (each cycle is 28 days)
  Time to Cmax (Tmax) of BBI-825 will be determined.
Area under the concentration time curve (AUC) of BBI-825 | Start of Cycle 1 until Day 1 of last treatment cycle (each cycle is 28 days)
  Area under the concentration time curve (AUC) of BBI-825 will be determined.
Anti-tumor activity of BBI-825 as determined by RECISTv1.1 | Start of Cycle 1 until Day 1 of last treatment cycle (each cycle is 28 days)
  Number of participants achieving a best response of progressive disease, stable disease, partial response, or complete response.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Doebele, MD, Study Director — Boundless Bio
Locations (5):
- United States (5):
  - Sarcoma Oncology Research Center, Santa Monica, California
  - START Midwest, Grand Rapids, Michigan
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - NEXT Oncology, Irving, Texas
  - NEXT Oncology, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No